CLINICAL TRIAL: NCT03263390
Title: Modeling the Neurological Basis and Characterizing the Neurological Phenotype of Obesity Using Human Neural Stem Cells
Status: Terminated | Type: Observational
Why Stopped: Study terminated by study partners
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Eduardo Grunvald, Clinical Professor of Medicine, University of California, San Diego
Other Study IDs: 170097
Record Dates: First submitted 2017-08-24; First posted 2017-08-28 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Obesity, Morbid
Keywords: Obesity; Bariatric Surgery; Anti Obesity Medications; Weight Regulation; Pluripotent Stem Cells
MeSH Terms: conditions — Obesity, Morbid; Obesity | interventions — Bariatric Surgery; Anti-Obesity Agents

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Fibroblasts, iPSCs, and DNA sequencing information generated from skin biopsies will be expanded and stored for potential future use.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Bariatric Surgery: Subjects that have demonstrated extreme response to bariatric surgery.
  Interventions: Procedure: Bariatric Surgery
- Anti Obesity Medications: Subjects that have demonstrated extreme response to anti obesity pharmacotherapy.
  Interventions: Drug: Anti Obesity Drugs

INTERVENTIONS:
Procedure: Bariatric Surgery — Sleeve gastrectomy or Roux-en-Y Gastric Bypass
  Groups: Bariatric Surgery
Drug: Anti Obesity Drugs — Response to FDA approved anti obesity medications
  Groups: Anti Obesity Medications

SUMMARY:
This study aims to characterize the neurological basis of obesity and response to surgical and medical treatment by inducing adult pluripotent stem cells into neuronal cells from subjects that have demonstrated extreme response to bariatric surgery or pharmacological treatment for obesity.

DETAILED DESCRIPTION:
The investigators will consent subjects who have achieved extreme response to either bariatric surgery or pharmacologic treatment for obesity and harvest fibroblasts from skin biopsies, which will be reprogrammed to induced pluripotent stem cells (iPSC). These iPSC's will then be differentiated into neural progenitor cells, neurons, astrocytes, and microglia to identify genetic and epigenetic pathways altered in disease-specific neural progenitor cells of the brain.

ELIGIBILITY:
Inclusion Criteria:

* History of obesity
* Treatment with bariatric surgery
* Treatment with anti obesity medications
* Greater than 70% excess weight loss at least 6 months after surgery
* Greater than 15% weight loss on anti obesity medications

Exclusion Criteria:

* Active cancer, not including non-melanoma skin cancer
* Active eating disorder
* Use of anti obesity medications in subjects with a history of bariatric surgery
* Active complication of the upper GI tract in patients with a history of bariatric surgery

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with obesity who are considered super responders to bariatric surgery or anti obesity pharmacotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2017-10-05 (Actual); Primary Completion 2020-08-10 (Actual); Study Completion 2020-08-10 (Actual)

PRIMARY OUTCOMES:
DNA sequencing | 4 months
  Perform DNA sequencing from skin biopsy progenitor cells
Generate human cell based models of obesity | 4 months
  Fibroblasts will be expanded in culture and then reprogrammed to hiPSCs.
Differentiation to human CNS cells | 4 months
  Disease specific hiPSCs cells will be differentiated into neural progenitor cells, neurons, astrocytes, and microglia
Identification of genetic and epigenetic pathways | 4 months
  Identify genetic and epigenetic pathways altered in disease-specific neural progenitor cells, neurons, and non-neuronal cells of the brain

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Grunvald, MD, Principal Investigator — UCSD
Locations (1):
- University of California San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No
This is not an intervention trial